CLINICAL TRIAL: NCT02770846
Title: Evaluation of Immediate Loading Versus Delayed Loading in Single-implant Restorations
Brief Title: Immediate Loading Versus Delayed Loading in Single-implant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Folktandvården Skåne AB (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RCT01BG; Dnr 2011/125 (Other: Regional Ethical Review Board in Lund)
Record Dates: First submitted 2016-04-26; First posted 2016-05-12 (Estimated); Results first posted 2020-03-26 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Immediate Dental Implant Loading
MeSH Terms: interventions — Immediate Dental Implant Loading

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate loading (Experimental): Immediate loading of single dental implant in the anterior maxilla with temporary crown in central occlusion
  Interventions: Procedure: Immediate loading
- Delayed loading (Active Comparator): Delayed loading. 2-stage procedure with a 4 months healing period before fabrication of temporary crown.
  Interventions: Procedure: Delayed loading

INTERVENTIONS:
Procedure: Immediate loading
  Arms: Immediate loading
Procedure: Delayed loading
  Arms: Delayed loading

SUMMARY:
The purpose of this prospective randomized clinical study was to compare implant survival, patient satisfaction, and radiographic, clinical, and aesthetic outcomes following immediate loading (IL) and delayed loading (DL) of single dental implants after 1,3 and 5 years of follow-up.

DETAILED DESCRIPTION:
Purpose: The objective of the present prospective randomized clinical study was to compare the overall treatment outcome following immediate loading (IL) and delayed loading (DL) of single implants after 5 year of follow-up.

Patients with a missing maxillary tooth (15-25) were randomly assigned to IL or DL. The protocol included implant installation in healed sites, immediate loading, delayed loading, temporary screw-retained restoration, and replacement with a permanent single implant crown. Outcome measures were implant survival, marginal bone level, soft tissue changes, papillae index, pink, and white esthetic score (PES and WES), patient judged aesthetics, and oral health impact profile (OHiP-14).

ELIGIBILITY:
Inclusion Criteria:

* Patients of at least 18 years of age.
* In need of one or more single-tooth replacements.
* The single-tooth replacement needs to be in the anterior maxilla
* Minimum of mesial-distal width of interdental space of 6 mm

Exclusion Criteria:

* General contraindications for oral surgery
* Inadequate oral hygiene
* Insufficient bone volume at the recipient site

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-04; Primary Completion 2015-12 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann Wennerberg, DDS, Phd, Study Director — Malmö University
Locations (1):
- Centre of Dental Specialist Care, Malmo, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Immediate Loading: Immediate loading of single dental implant in the anterior maxilla with temporary crown in central occlusion
  Immediate loading
- Delayed Loading: Delayed loading. 2-stage procedure with a 4 months healing period before fabrication of temporary crown.
  Delayed loading
Period: Overall Study
Arm/Group | Immediate Loading | Delayed Loading
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Immediate Loading: Immediate loading with a screw-retained temporary crown and replacement with a permanent crown.
- Delayed Loading: Delayed loading with a temporary crown to optimize the emergence profile and replacement with a permanent crown.
- Total: Total of all reporting groups
Arm/Group | Immediate Loading | Delayed Loading | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.8 (13.3) | 40.9 (15.5) | 40.9 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 19 | 30
  Male | 14 | 6 | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Level of Marginal Bone
Description: Digital intra-oral periapical radiographs at different time points. The marginal bone level is measured after calibration. Measurements are taken from the implant-abutment junction to the marginal bone level (millimetres). Change in marginal bone level is calculated by comparing bone-to-implant contact level of all appointments to radiographic baseline.
Time Frame: Baseline to 12 months
Population: In the delayed group 1 implant was lost prior to evaluation and therefore not possible to include in this evaluation. Reported as a serious event.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Immediate Loading | Delayed Loading
Number analyzed (Participants) | 25 | 24
mm | -0.57 (0.52) | -0.69 (0.69)

2. Primary Outcome: Pink Esthetic Score
Description: The Pink esthetic score (PES) measures the aesthetic appearance of mucosa tissue at the implant site.
  Intraoral photographs from the aesthetic baseline and follow-up appointments are used to register the pink esthetic score, an objective aesthetic scale were the shape,size,colour and structure of the soft tissue is rated.
  The scale consists of 7 variables that are scored 0,1 or 2, the 7 variables scores are combined.
  Scale range 0-14, 0 minimum and 14 maximum. A higher score represent a better aesthetic outcome.
Time Frame: After 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Immediate Loading | Delayed Loading
Number analyzed (Participants) | 25 | 24
units on a scale | 10.36 (2.46) | 10.67 (2.32)

3. Primary Outcome: Oral Health Impact Profile 14
Description: The Oral Health Impact Profile 14 (OHIP-14) measure oral health related quality of life.
  The oral health-related quality of life is calculated using the Swedish validated version of the Oral Health Impact Profile (OHIP-14) questionnaire. The questionnaires are completed at the beginning of the treatment and 12 months after the definitive crown placement.
  The scale consists of 14 variables that are scored 1,2,3,4 or 5, the 14 variables scores are combined.
  Scale range 14-70, 14 minimum and 70 maximum. A low score represent a better oral health related quality of life.
Time Frame: Pre-surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Immediate Loading | Delayed Loading
Number analyzed (Participants) | 25 | 25
units on a scale | 26.68 (9.3) | 23.40 (8.64)

4. Primary Outcome: White Esthetic Score
Description: The White esthetic score (WES) measures the aesthetic appearance of the implant crown.
  Intraoral photographs from the aesthetic baseline and follow-up appointments are used to register the white esthetic score, an objective aesthetic scale were the shape,size,colour and structure of the implant crown is rated.
  The scale consists of 5 variables that are scored 0,1 or 2, the 5 variables scores are combined.
  Scale range 0-10, 0 minimum and 10 maximum. A higher score represent a better aesthetic outcome.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Immediate Loading | Delayed Loading
Number analyzed (Participants) | 25 | 24
units on a scale | 7.00 (1.41) | 7.00 (1.64)

5. Primary Outcome: Pink Esthetic Score
Description: as for outcome 2
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Loading | Delayed Loading
Number analyzed (Participants) | 25 | 24
score on a scale | 8.56 (2.27) | 9.42 (2.98)

6. Primary Outcome: Oral Health Impact Profile 14 (OHIP-14)
Description: as for outcome 3
Time Frame: After 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Immediate Loading | Delayed Loading
Number analyzed (Participants) | 25 | 24
units on a scale | 16.48 (3.87) | 15.38 (2.58)

7. Primary Outcome: White Esthetic Score
Description: as for outcome 4
Time Frame: After 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Immediate Loading | Delayed Loading
Number analyzed (Participants) | 25 | 24
Score on a scale | 7.76 (1.30) | 7.87 (1.39)

8. Primary Outcome: Change in Level of Marginal Bone
Description: as for outcome 1
Time Frame: Baseline to 5 years
Population: In the delayed group 1 implant was lost prior to evaluation and therefore not possible to include in this evaluation. Reported as a serious event.
  1 patient was lost to follow-up in the immediate loading group and 1 in the delayed loading group.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Immediate Loading | Delayed Loading
Number analyzed (Participants) | 24 | 23
mm | -0.50 (0.73) | -0.54 (0.65)

9. Primary Outcome: Pink Esthetic Score
Description: as for outcome 2
Time Frame: After 5 year
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Immediate Loading | Delayed Loading
Number analyzed (Participants) | 24 | 23
Score on a scale | 11.00 (2.08) | 11.17 (2.39)

10. Primary Outcome: White Esthetic Score
Description: as for outcome 4
Time Frame: 5 years
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Immediate Loading | Delayed Loading
Number analyzed (Participants) | 24 | 23
Score on a scale | 7.63 (1.53) | 7.91 (1.53)

ADVERSE EVENTS:
Time Frame: 1 year
Description: Serious events: loss of dental implant. Other adverse event: prosthetic restoration complications.
Arm/Group | Immediate Loading | Delayed Loading
Serious Adverse Events (participants affected / at risk) | 0/25 | 1/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immediate Loading (N=25) | Delayed Loading (N=25)
Dental implant loss (Surgical and medical procedures) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes